CLINICAL TRIAL: NCT00960934
Title: A Phase IIb, Randomized, Placebo-Controlled, Dose-Ranging Study of MK-5442 in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: A Dose-Ranging Study of MK-5442 in Postmenopausal Women With Osteoporosis (MK-5442-001)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5442-001; 2009-012926-35 (EudraCT Number)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Postmenopausal; MK-5442
MeSH Terms: conditions — Osteoporosis | interventions — JTT 305; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK-5442 2.5 mg (Experimental): Following a 2-week open-label placebo run-in, participants received a daily oral dose of 2.5 mg of MK-5442 for a duration of at least 6 months.
  Interventions: Drug: MK-5442; Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- MK-5442 5 mg (Experimental): Following a 2-week open-label placebo run-in, participants received a daily oral dose of 5 mg of MK-5442 for a duration of at least 6 months.
  Interventions: Drug: MK-5442; Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- MK-5442 7.5 mg (Experimental): Following a 2-week open-label placebo run-in, participants received a daily oral dose of 7.5 mg of MK-5442 for a duration of at least 6 months.
  Interventions: Drug: MK-5442; Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- MK-5442 10 mg (Experimental): Following a 2-week open-label placebo run-in, participants received a daily oral dose of 10 mg of MK-5442 for a duration of at least 6 months.
  Interventions: Drug: MK-5442; Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- MK-5442 15 mg (Experimental): Following a 2-week open-label placebo run-in, participants received a daily oral dose of 15 mg of MK-5442 for a duration of at least 6 months.
  Interventions: Drug: MK-5442; Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Placebo (Placebo Comparator): Following a 2-week open-label placebo run-in, participants received a daily oral dose of placebo dose-matched to MK-5442 for a duration of at least 6 months.
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: MK-5442 — MK-5442 2.5 mg, 5 mg, 7.5 mg, 10 mg, or 15 mg tablet once daily for at least 6 months.
  Arms: MK-5442 10 mg; MK-5442 15 mg; MK-5442 2.5 mg; MK-5442 5 mg; MK-5442 7.5 mg
Drug: Placebo — Dose-matched oral placebo to MK-5442
Dietary Supplement: Vitamin D3 — Vitamin D3, two 400 IU tablets daily throughout the study.
Dietary Supplement: Calcium carbonate — Participants who had a calcium intake of less than 1200 mg/day at baseline received a daily 500 mg calcium supplement throughout the study.

SUMMARY:
The purpose of this study was to identify an appropriate dose of

MK-5442 that produced an osteoanabolic effect without causing hypercalcemia in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
Amendment 4 of the protocol changed the duration of the study from 2 years to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for at least 5 years
* No history of fragility fracture, unless participant is not willing to take marketed osteoporosis therapy or is not a candidate for marketed osteoporosis therapy
* Agrees not to use medications for osteoporosis except medications associated with the study
* Areal bone mineral density (BMD) T-score <-2.5 at one or more of the following 4 BMD sites: total hip, femoral neck, trochanter, or lumbar spine and is ≥ -3.5 at all 4 BMD sites. Participants unwilling to take or ineligible for marketed osteoporosis therapy may have one or more areal BMD T-scores of < -3.5

Exclusion Criteria:

* Unable to undergo dual-energy X-ray absorptiometry (DXA) scan due to obesity (ie, weight >250 lbs)
* Use of oral bisphosphonates in the 6 months prior to study screening, for more than 3 months in the past 2 years, or lifetime use of more than 6 months
* Use of intravenous bisphosphonates, strontium, or growth hormone at any time
* Use of phenytoin or heparin within 2 weeks prior to Visit 1; use of raloxifene within 6 months prior to Visit 1
* Use of pioglitazone or rosiglitazone at study screening
* Use of estrogen ± progestin, in any form other than vaginal or topical application, for 6 months prior to Study Visit 1
* Prior total thyroidectomy
* Human immunodeficiency virus (HIV)- positive or acquired immune deficiency syndrome (AIDS)-related illness
* History of malignant cancer within 5 years of study screening, except for certain skin or cervical cancers
* History of Paget's disease and/or kidney stones
* An active user of any illicit drug
* History of or active alcohol abuse
* Participated in an investigational drug study within the past 30 days

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

REFERENCES:
- [Result] Halse J, Greenspan S, Cosman F, Ellis G, Santora A, Leung A, Heyden N, Samanta S, Doleckyj S, Rosenberg E, Denker AE. A phase 2, randomized, placebo-controlled, dose-ranging study of the calcium-sensing receptor antagonist MK-5442 in the treatment of postmenopausal women with osteoporosis. J Clin Endocrinol Metab. 2014 Nov;99(11):E2207-15. doi: 10.1210/jc.2013-4009. Epub 2014 Aug 28. PMID 25166719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 383 participants were randomized on study and 380 participants were treated on study.
Period: Overall Study
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Started | 64 | 63 | 64 | 64 | 64 | 64
Number Treated | 64 | 62 (1 participant was randomized but not treated) | 64 | 64 | 63 (1 participant was randomized but not treated) | 63 (1 participant was randomized but not treated)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 64 | 63 | 64 | 64 | 64 | 64
Not completed — Adverse Event | 2 | 3 | 3 | 2 | 4 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 5 | 4 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 1 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 4 | 0 | 3 | 3 | 2
Not completed — Withdrawal by Subject | 5 | 6 | 4 | 5 | 5 | 7
Not completed — Study Terminated by Sponsor | 50 | 46 | 52 | 50 | 49 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 64 | 64 | 64 | 64 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (6.3) | 67.3 (6.5) | 67.4 (6.0) | 67.8 (6.4) | 66.5 (5.4) | 67.6 (6.7) | 67.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 64 | 64 | 64 | 64 | 383
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Percent Change From Baseline to Month 6 in Lumbar Spine Areal Bone Mineral Density (aBMD)
Description: Dual Energy X-ray Absorptiometry (DXA) was used to assess and measure aBMD of the lumbar spine. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline (BL) and Month 6
Population: Full Analysis Set (FAS); participants who received at least one dose of study treatment, had post-randomization data subsequent to at least one dose of study treatment, and who had baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 58 | 54 | 56 | 55 | 56 | 56
percent change | 0.74 [-0.21 to 1.68] | 1.50 [0.53 to 2.48] | 0.92 [-0.02 to 1.87] | 1.69 [0.73 to 2.64] | 1.13 [0.18 to 2.08] | 0.57 [-0.40 to 1.55]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.749, Longitudinal Data Analysis Model — The Type-I error rate over the multiple treatment dose comparisons for the areal BMD at lumbar spine endpoint were controlled by step-down Dunnett's test at the primary time point of Month 6, at an alpha level of 0.05, two-sided; LS Mean Difference in Change From BL = 0.56, 95% CI 2-sided [-1.04 to 2.16]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.333, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference in Change From BL = 1.12, 95% CI 2-sided [-0.60 to 2.83]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.823, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference in Change From BL = 0.35, 95% CI 2-sided [-1.14 to 1.84]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.457, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference in Change From BL = 0.93, 95% CI 2-sided [-0.75 to 2.61]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.823, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference in Change From BL = 0.16, 95% CI 2-sided [-1.17 to 1.50]

2. Primary Outcome: Percentage of Participants With Total Serum Calcium Levels Outside the Pre-defined Limits of Change
Description: Normal serum calcium level is 8-10 mg/dL (2-2.5 mmol/L) with some interlaboratory variation in the reference range, and hypercalcemia is defined as a serum calcium level greater than 10.5 mg/dL (>2.5 mmol/L).
  Based on these references, ≥10.6 mg/dL was predefined in this study as the cut-off for the normal limits of change. Participants with calcium levels ≥10.6 mg/dL were considered as having a "Tier 1" safety event.
Time Frame: Baseline through Month 6
Population: All Participants as Treated (APaT) population; all randomized participants who received at least one dose of study treatment. 3 randomized participants did not receive treatment and were not included in the APaT.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 64 | 62 | 64 | 64 | 63 | 63
Percentage of participants | 7.8 | 32.3 | 32.8 | 56.3 | 73.0 | 3.2
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; The Miettinen and Nurminen Method was used to estimate the treatment differences between the active dose group and the placebo group by comparing the percentage of participants in the active dose group with the event vs. the percentage of participants in the placebo group with the event. An associated p-value and 95% confidence interval were calculated for this difference; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 69.8, 95% CI [56.5 to 80.0]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 53.1, 95% CI 2-sided [39.6 to 65.2]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 29.6, 95% CI 2-sided [17.6 to 42.4]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 29.1, 95% CI 2-sided [17.0 to 42.0]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.254, Miettinen and Nurminen Method; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-4.1 to 14.4]

3. Primary Outcome: Percentage of Participants With Albumin-Corrected Calcium Levels Outside the Pre-defined Limits of Change
Description: Albumin-Corrected Calcium = ([4 - plasma albumin in g/dL] × 0.8 + serum calcium).
  ≥10.6 mg/dL was predefined in this study as the cut-off for the normal limits of change. Participants with albumin-corrected calcium levels ≥10.6 mg/dL were considered as having a "Tier 1" safety event.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 64 | 62 | 64 | 64 | 63 | 63
Percentage of participants | 0.0 | 9.7 [2.96 to 5.35] | 18.8 [2.75 to 5.09] | 37.5 [4.28 to 6.69] | 49.2 [5.10 to 7.50] | 1.6 [-1.04 to 1.22]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 47.6, 95% CI 2-sided [34.9 to 60.0]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 35.9, 95% CI 2-sided [24.1 to 48.5]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, Miettinen and Nurminen Method; Mean Difference (Final Values) = 17.2, 95% CI 2-sided [7.7 to 28.7]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.050, Miettinen and Nurminen Method; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [-0.0 to 18.2]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.313, Miettinen and Nurminen Method; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-8.5 to 4.2]

4. Primary Outcome: Percentage of Participants With Kidney Stones
Description: Evidence of kidney stone(s) was considered an event of interest and was prespecified as a "Tier 1" safety event.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 64 | 62 | 64 | 64 | 63 | 63
Percentage of participants | 1.6 | 1.6 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen Method; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-5.8 to 5.8]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen Method; Mean Difference (Final Values) = 0, 95% CI 2-sided [-5.8 to 5.7]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen Method; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-5.8 to 5.7]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.313, Miettinen and Nurminen Method; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-4.2 to 8.6]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.321, Miettinen and Nurminen Method; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-4.3 to 8.4]

5. Primary Outcome: Percentage of Participants With Bone Neoplasms
Description: Evidence of bone neoplasm(s) was considered an event of interest and was prespecified as a "Tier 1" safety event.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 64 | 62 | 64 | 64 | 63 | 63
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Total Hip aBMD
Description: DXA was used to assess and measure aBMD of the total hip. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 58 | 54 | 56 | 55 | 56 | 56
percent change | -0.20 [-0.95 to 0.55] | -0.32 [-1.10 to 0.46] | 0.32 [-0.43 to 1.07] | 0.07 [-0.69 to 0.82] | 0.33 [-0.43 to 1.08] | 0.08 [-0.69 to 0.86]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.959, Longitudinal Data Analysis Model — The Type-I error rate over the multiple treatment dose comparisons were controlled by step-down Dunnett's test at the primary time point of Month 6, at an alpha level of 0.05, two-sided; LS Mean Difference in Change From BL = 0.24, 95% CI 2-sided [-1.03 to 1.51]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.971, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.02, 95% CI 2-sided [-1.08 to 1.04]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.959, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.24, 95% CI 2-sided [-0.95 to 1.42]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.915, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.41, 95% CI 2-sided [-1.78 to 0.97]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.959, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.28, 95% CI 2-sided [-1.60 to 1.04]

7. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Femoral Neck aBMD
Description: DXA was used to assess and measure aBMD of the femoral neck. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 58 | 54 | 56 | 55 | 56 | 56
percent change | 1.23 [0.21 to 2.25] | -0.52 [-1.58 to 0.54] | 0.12 [-0.89 to 1.14] | -0.20 [-1.23 to 0.83] | 0.54 [-0.48 to 1.56] | -0.04 [-1.09 to 1.01]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.849, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.58, 95% CI 2-sided [-1.22 to 2.37]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.964, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.16, 95% CI 2-sided [-1.79 to 1.47]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.964, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.16, 95% CI 2-sided [-1.27 to 1.59]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.855, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.48, 95% CI 2-sided [-2.23 to 1.27]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.287, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 1.27, 95% CI 2-sided [-0.58 to 3.12]

8. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Trochanter aBMD
Description: DXA was used to assess and measure aBMD of the trochanter. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 58 | 54 | 56 | 55 | 56 | 56
percent change | 0.41 [-0.78 to 1.60] | 0.95 [-0.29 to 2.19] | 0.54 [-0.65 to 1.74] | 0.49 [-0.72 to 1.70] | 1.10 [-0.11 to 2.30] | 0.49 [-0.74 to 1.73]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.933, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.60, 95% CI 2-sided [-1.56 to 2.77]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.999, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.01, 95% CI 2-sided [-1.69 to 1.68]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.999, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.05, 95% CI 2-sided [-1.84 to 1.93]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.959, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.45, 95% CI 2-sided [-1.67 to 2.57]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.999, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.08, 95% CI 2-sided [-2.10 to 1.94]

9. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Total Body aBMD
Description: DXA was used to assess and measure aBMD of the total body. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 51 | 51 | 54 | 50 | 53 | 52
percent change | 0.43 [-0.11 to 0.97] | 0.28 [-0.28 to 0.84] | 0.80 [0.27 to 1.33] | 0.21 [-0.35 to 0.76] | 0.09 [-0.44 to 0.63] | 0.27 [-0.29 to 0.82]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.976, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.17, 95% CI 2-sided [-1.12 to 0.77]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.982, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.06, 95% CI 2-sided [-0.93 to 0.80]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.489, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.53, 95% CI 2-sided [-0.43 to 1.49]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.982, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.02, 95% CI 2-sided [-0.75 to 0.78]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.976, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.16, 95% CI 2-sided [-0.76 to 1.08]

10. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Distal One-third Forearm Areal BMD
Description: DXA was used to assess and measure aBMD of the distal 1/3 forearm. Areal BMD was measured as "areal" density using units of gram (gm) of tissue /centimeter of tissue squared (cm^2).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 51 | 51 | 55 | 49 | 53 | 52
percent change | -0.47 [-1.42 to 0.48] | -0.32 [-1.30 to 0.65] | 0.44 [-0.47 to 1.36] | -0.49 [-1.46 to 0.48] | -0.56 [-1.50 to 0.37] | -0.21 [-1.18 to 0.76]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.961, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.35, 95% CI 2-sided [-2.00 to 1.31]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.961, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.28, 95% CI 2-sided [-1.90 to 1.34]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.778, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.66, 95% CI 2-sided [-1.01 to 2.33]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.961, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.11, 95% CI 2-sided [-1.45 to 1.24]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.961, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.25, 95% CI 2-sided [-1.77 to 1.26]

11. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Trabecular Volumetric BMD of the Hip
Description: Quantitative computed tomography (QCT) technology was used to assess and measure bone mineral content volumetrically (ie, in grams of tissue per centimeter of tissue cubed).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 42 | 43 | 46 | 39 | 41 | 50
percent change | -0.41 [-1.44 to 0.62] | -0.34 [-1.43 to 0.75] | -0.89 [-1.90 to 0.13] | -0.88 [-1.97 to 0.22] | -0.80 [-1.87 to 0.26] | -0.37 [-1.37 to 0.63]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.901, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.43, 95% CI 2-sided [-2.03 to 1.17]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.901, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.51, 95% CI 2-sided [-2.18 to 1.17]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.901, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.52, 95% CI 2-sided [-2.17 to 1.13]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.997, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.03, 95% CI 2-sided [-1.29 to 1.35]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.997, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.04, 95% CI 2-sided [-1.51 to 1.43]

12. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Trabecular Volumetric BMD of the Lumbar Spine
Description: Quantitative computed tomography (QCT) technology was used at baseline and periodically through out the study to assess and measure bone mineral content volumetrically (ie, in grams of tissue per centimeter of tissue cubed).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 43 | 43 | 44 | 39 | 40 | 50
percent change | 1.94 [0.13 to 3.75] | 0.94 [-0.97 to 2.85] | 1.83 [0.02 to 3.64] | 3.35 [1.43 to 5.27] | 1.06 [-0.83 to 2.96] | 1.43 [-0.33 to 3.19]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.979, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.37, 95% CI 2-sided [-2.73 to 1.99]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.363, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 1.92, 95% CI 2-sided [-1.10 to 4.95]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.979, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.40, 95% CI 2-sided [-2.18 to 2.98]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.979, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.49, 95% CI 2-sided [-3.27 to 2.30]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.979, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 0.51, 95% CI 2-sided [-2.34 to 3.37]

13. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in the Ratio of Urinary N-Telopeptides of Type I Collagen to Creatinine (u-NTx/Cr)
Description: The ratio of u-NTx to Cr is a biomarker for bone resorption. It is measured in the serum in units of nanomoles (nm) of bone collagen equivalents (BCE)/millimoles of creatinine (Cr).
Time Frame: Baseline and Month 6
Population: Per Protocol population; defined as the subset of the APaT population that excluded participants based on critical protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 50 | 51 | 53 | 51 | 52 | 53
percent change | -12.18 [-21.23 to -2.10] | -9.46 [-18.87 to 1.03] | -20.73 [-28.79 to -11.76] | -7.82 [-17.33 to 2.78] | 1.87 [-8.53 to 13.45] | -17.90 [-26.15 to -8.73]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p = 0.020, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 19.77, 95% CI 2-sided [2.26 to 37.46]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.357, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 10.08, 95% CI 2-sided [-6.16 to 26.41]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.642, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -2.83, 95% CI 2-sided [-14.81 to 9.14]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.434, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 8.44, 95% CI 2-sided [-7.09 to 24.04]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.579, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 5.72, 95% CI [-8.62 to 20.10]

14. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Serum C-Terminal Telopeptide Collagen I (s-CTx)
Description: C-Terminal Telopeptide Collagen I is used as a serum-marker of bone resorption in the assessment of osteoporosis.
Time Frame: Baseline to Month 6
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 54 | 52 | 52 | 52
percent change | -15.39 [-23.80 to -6.05] | -5.87 [-15.32 to 4.63] | -4.93 [-14.23 to 5.39] | 5.68 [-4.77 to 17.27] | 19.37 [7.60 to 32.43] | -14.89 [-23.24 to -5.64]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 34.26, 95% CI 2-sided [15.27 to 53.56]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p = 0.014, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 20.57, 95% CI 2-sided [3.28 to 38.02]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.307, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 9.97, 95% CI 2-sided [-5.69 to 25.70]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.307, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 9.02, 95% CI 2-sided [-5.85 to 23.95]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.937, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = -0.50, 95% CI 2-sided [-12.92 to 11.92]

15. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Serum Bone-Specific Alkaline Phosphatase (s-BSAP)
Description: Bone Specific Alkaline Phosphatase is a biomarker of bone formation and is measured in units of microgram (μg)/liter (L).
Time Frame: Baseline and Month 6
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 54 | 52 | 52 | 52
percent change | -0.60 [-6.87 to 6.10] | 0.26 [-6.17 to 7.13] | 4.39 [-2.13 to 11.35] | 17.33 [9.93 to 25.22] | 13.13 [6.02 to 20.72] | -6.05 [-11.92 to 0.20]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 19.19, 95% CI 2-sided [7.42 to 31.02]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 23.38, 95% CI 2-sided [11.02 to 35.82]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.061, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 10.45, 95% CI 2-sided [-0.37 to 21.30]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.283, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 6.31, 95% CI 2-sided [-3.81 to 16.45]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.283, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 5.46, 95% CI 2-sided [-3.39 to 14.31]

16. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Serum Procollagen Type I N-Terminal Propeptide (P1NP)
Description: Measurement of P1NP appears to be a sensitive marker of bone formation rate in the assessment of osteoporosis.
Time Frame: Baseline to Month 6
Population: The 'Per Protocol' population was used for this analysis. The Per-Protocol population was defined as a subset population that excluded participants based on critical protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 54 | 52 | 52 | 52
percent change | -9.97 [-18.46 to -0.59] | -9.76 [-18.36 to -0.26] | 2.33 [-7.16 to 12.78] | 21.30 [9.91 to 33.88] | 38.41 [25.45 to 52.71] | -18.36 [-25.96 to -9.97]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p < .001, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 56.77, 95% CI 2-sided [37.62 to 76.35]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p < .001, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 39.66, 95% CI 2-sided [22.44 to 57.17]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p = 0.003, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 20.68, 95% CI 2-sided [5.72 to 35.78]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.265, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 8.59, 95% CI 2-sided [-4.81 to 22.05]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.265, Longitudinal Data Analysis — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 8.39, 95% CI 2-sided [-3.40 to 20.21]

17. Secondary Outcome: LS Mean Percent Change From Baseline to Month 6 in Serum Osteocalcin
Description: Serum osteocalcin is a biomarker of bone formation and is measured using units of nanograms (ng) / milliliter (mL).
Time Frame: Baseline and Month 6
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 54 | 52 | 52 | 52
percent change | -11.61 [-18.19 to -4.50] | -2.75 [-10.10 to 5.19] | 9.18 [1.15 to 17.86] | 25.79 [16.45 to 35.88] | 37.43 [27.24 to 48.42] | -15.62 [-21.83 to -8.92]
Statistical Analysis 1: Comparison: MK-5442 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 53.05, 95% CI 2-sided [37.83 to 68.53]
Statistical Analysis 2: Comparison: MK-5442 10 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 41.41, 95% CI 2-sided [27.36 to 55.65]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 24.81, 95% CI 2-sided [12.39 to 37.33]
Statistical Analysis 4: Comparison: MK-5442 5 mg vs Placebo; Test type: Superiority or Other; p = 0.020, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 12.87, 95% CI 2-sided [1.73 to 24.06]
Statistical Analysis 5: Comparison: MK-5442 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.397, Longitudinal Data Analysis Model — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference in Change From BL = 4.02, 95% CI 2-sided [-5.31 to 13.36]

ADVERSE EVENTS:
Time Frame: From October 2, 2009 to December 21, 2010, with an in-house data-cut date of February 10, 2011
Description: All Participants as Treated (APaT) Population. Three participants were randomized but not treated, and thus are not included in the adverse event table calculations (one participant was randomized to 5 mg MK-5442; one participant was randomized to 15 mg MK-5442 and one participant was randomized to Placebo.
Arm/Group | MK-5442 2.5 mg | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/64 | 0/62 | 4/64 | 5/64 | 4/63 | 3/63
Other Adverse Events (participants affected / at risk) | 18/64 | 24/62 | 15/64 | 28/64 | 18/63 | 26/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5442 2.5 mg (N=64) | MK-5442 5 mg (N=62) | MK-5442 7.5 mg (N=64) | MK-5442 10 mg (N=64) | MK-5442 15 mg (N=63) | Placebo (N=63)
Angina pectoris aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary stent stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postural hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5442 2.5 mg (N=64) | MK-5442 5 mg (N=62) | MK-5442 7.5 mg (N=64) | MK-5442 10 mg (N=64) | MK-5442 15 mg (N=63) | Placebo (N=63)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 7 (7) | 5 (5) | 4 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 5 (5)
Tiredness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Chest Infection (Infections and infestations) | 2 (2) | 1 (2) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Common Cold (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 3 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 6 (7)
Urinary Tract Infection (Infections and infestations) | 5 (8) | 5 (6) | 2 (3) | 10 (12) | 3 (5) | 6 (6)
Pain in Hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 2 (3) | 4 (4) | 5 (5) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator and/or his/her colleagues may publish the results of the study associated with their study site independently.